CLINICAL TRIAL: NCT05276505
Title: Evaluation of the Efficacy of Two Different Aromatherapy Methods in Reducing Anxiety Before Breast Biopsy
Brief Title: Aromatherapy Methods in Reducing Anxiety Before Breast Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Acibadem University, Asisst. Prof., Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK 2021-14/18
Record Dates: First submitted 2022-03-03; First posted 2022-03-11 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2021-07

CONDITIONS: Patient Relations, Nurse; Patient Satisfaction; Anxiety State; Breast Cancer
Keywords: breast cancer; aromatherapy; anxiety
MeSH Terms: conditions — Patient Satisfaction; Anxiety Disorders; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group - Standardized care (No Intervention): Standardized nursing care applications
  Evaluation with STAI scale (anxiety levels) breast biopsy Evaluation with the STAI scale (anxiety levels) after the breast biopsy procedure
- Experimental Group- Lavender Aromatherapy Tablet (Experimental): Before 20 minutes from breast biopsy. Lavender aromatherapy tablets. A small (approximately 1x 0.5 inch), rectangular, absorbent tablet containing 2 ml of lavender essential oil (10) was adhered to the patient's shoulder level in the waiting room.
  Patients were asked to inhale the aromatherapy tablet for 20 minutes before the procedure.
  Evaluation with STAI scale (anxiety levels) breast biopsy Evaluation with the STAI scale (anxiety levels) after the breast biopsy procedure
  Interventions: Other: Lavender Aromatherapy Tablet
- Experimental Group- Lavender-Mint Aromatherapy Tablet (Experimental): Before 20 minutes from breast biopsy. Lavender-Mint aromatherapy tablets. A small (approximately 1x 0.5 inch), rectangular, absorbent tablet containing 2 ml of lavender essential oil (10) was adhered to the patient's shoulder level in the waiting room.
  Patients were asked to inhale the aromatherapy tablet for 20 minutes before the procedure.
  Evaluation with STAI scale (anxiety levels) breast biopsy Evaluation with the STAI scale (anxiety levels) after the breast biopsy procedure
  Interventions: Other: Lavender Aromatherapy Tablet

INTERVENTIONS:
Other: Lavender Aromatherapy Tablet — Before the breast biopsy, aromatherapy tablets was adhered to the patient's shoulder in the waiting room and were asked to sniff
  Other Names: Lavender-Mint Aromatherapy Tablet
  Arms: Experimental Group- Lavender Aromatherapy Tablet; Experimental Group- Lavender-Mint Aromatherapy Tablet

SUMMARY:
A breast biopsy is a cause for anxiety for most women when faced with a diagnosis of breast cancer. Physiological and psychological effects of breast biopsy may continue in the pre-biopsy and post-biopsy period. The aim of this study is to compare the effectiveness of two different aromatherapy methods applied in reducing anxiety before breast biopsy.

DETAILED DESCRIPTION:
Anxiety level was evaluated according to objective criteria by pretesting and posttesting lavender, lavender-mint and odorless (placebo) aromatherapy tablets applied before the biopsy in patients scheduled for breast biopsy.

The study was conducted with 135 patients, 90 of whom were in the experimental group and 45 in the control group. Patients were randomly assigned to the experimental and control groups according to their sequence numbers.

Before the biopsy, lavender aromatherapy and lavender-mint aromatherapy tablets were administered to the experimental group, and an odorless (placebo) aromatherapy tablet to the control group. Aromatherapy tablets 20 minutes after the procedure. First, a small (approximately 1x 0.5 inch), rectangular, absorbent, self-adhesive tablet containing 2 ml of lavender essential oil (10) was adhered to the patient's shoulder level. Research data were collected with the "Spielberger State Anxiety Scale" to determine the level of anxiety before and after breast biopsy.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* Female patients scheduled for breast biopsy (stereotactic biopsy, ultrasound biopsy, magnetic resonance imaging biopsy)
* Individuals who can speak, understand and communicate in Turkish will be included in the study.

Exclusion Criteria:

* Pregnant and lactating women,
* Patients who are allergic to plants (lavender/lavender-mint),
* Patients with a diagnosis of psychiatric illness, migraine, chronic headache or sense of smell
* Patients who have difficulty breathing through their nose
* People who can't smell, who are sensitive to smells or smells
* Patients with a history of asthma, epilepsy or seizures as a precaution.
* Patients with active wheezing
* Patients with cognitive, verbal or hearing problems that may affect communication

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
State Anxiety Level | Evaluation of the differences between anxiety scales score - The scale is filled in 2 times - before breast biopsy (1), and after immediately breast biopsy (2)
  State Anxiety Level is evaluated by Spielberger State-Trait Anxiety Inventory - This inventory is a four-degree Likert type scale ranging from "Almost never" to "Almost always". In the state anxiety scale, the individual evaluates how he/ she feels "right now". The total score obtained from each scale varies between 20 and 80. A high score indicates a high anxiety level, a low score indicates a low anxiety level

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Uslu, Asisst Prof, Study Director — Acıbadem Üniversitesi
Locations (1):
- Yasemin Uslu, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Trambert R, Kowalski MO, Wu B, Mehta N, Friedman P. A Randomized Controlled Trial Provides Evidence to Support Aromatherapy to Minimize Anxiety in Women Undergoing Breast Biopsy. Worldviews Evid Based Nurs. 2017 Oct;14(5):394-402. doi: 10.1111/wvn.12229. Epub 2017 Apr 10. PMID 28395396
- [Result] Franco L, Blanck TJ, Dugan K, Kline R, Shanmugam G, Galotti A, von Bergen Granell A, Wajda M. Both lavender fleur oil and unscented oil aromatherapy reduce preoperative anxiety in breast surgery patients: a randomized trial. J Clin Anesth. 2016 Sep;33:243-9. doi: 10.1016/j.jclinane.2016.02.032. Epub 2016 May 5. PMID 27555173
- [Result] Tola YO, Chow KM, Liang W. Effects of non-pharmacological interventions on preoperative anxiety and postoperative pain in patients undergoing breast cancer surgery: A systematic review. J Clin Nurs. 2021 Dec;30(23-24):3369-3384. doi: 10.1111/jocn.15827. Epub 2021 May 3. PMID 33942405
- [Result] Beyliklioglu A, Arslan S. Effect of Lavender Oil on the Anxiety of Patients Before Breast Surgery. J Perianesth Nurs. 2019 Jun;34(3):587-593. doi: 10.1016/j.jopan.2018.10.002. Epub 2019 Jan 16. PMID 30660371
- [Result] Jaruzel CB, Gregoski M, Mueller M, Faircloth A, Kelechi T. Aromatherapy for Preoperative Anxiety: A Pilot Study. J Perianesth Nurs. 2019 Apr;34(2):259-264. doi: 10.1016/j.jopan.2018.05.007. Epub 2018 Sep 8. PMID 30205934